CLINICAL TRIAL: NCT07389642
Title: Management of Patients With Brain-onset Oligometastatic Non-small-cell Lung Cancer (NSCLC)
Brief Title: Brain Oligometastasis in NSCLC
Acronym: OligoLung
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2025/058
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Brain Oligometastatic; Non-small Cell Lung Cancer
Keywords: Metastatic NSCLC; Brain metastasis; Oligometastasis; Survival
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Local treatments: Local multimodal treatments (thoracic surgery/radiotherapy + brain surgery/radiotherapy)
  Interventions: Other: Standard treatments / multiple strategies
- Systemic treatment: Chemoimmunotherapy combination
  Interventions: Other: Standard treatments / multiple strategies

INTERVENTIONS:
Other: Standard treatments / multiple strategies — Standard treatments / multiple strategies

SUMMARY:
75-80% of NSCLC are diagnosed at the metastatic stage. Among the most frequent sites are brain metastases. The management of patients with exclusive limited brain involvement is not standardized. The question is therefore which therapeutic strategy is optimal in such disease presentation. We will analyze the impact of different therapeutic strategies on patients treated at Bordeaux University Hospital and the Bergonié Institute

DETAILED DESCRIPTION:
75-80% of NSCLC are diagnosed at the metastatic stage. Among the most frequent sites are brain metastases. The management of patients with exclusive limited brain involvement is not standardized. The question is therefore which therapeutic strategy is optimal in terms of disease control: local treatment of the main tumor and brain versus systemic treatment with chemotherapy and immunotherapy. We will analyze the impact of these 2 strategies on patients treated at Bordeaux University Hospital and the Bergonié Institute.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients managed at Bordeaux University Hospital
* Non-small-cell lung cancer
* Oligometastatic brain cancer (fewer than 5 lesions at diagnosis)
* Patient over 18 years old

Exclusion Criteria:

* Oncogenic addiction EGFR, ALK, ROS1
* Patient with concomitant cancer
* Patient with prior treatment for lung cancer in the year preceding diagnosis at metastatic stage

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patient with NSCLC treated at CHU Bordeaux and Bergonié Institute
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Once, at progression or death from any cause
  Time from random assignment in a clinical trial to disease progression or death from any cause

SECONDARY OUTCOMES:
PFS from the date of the next treatment to disease progression or death from any cause (PFS2) | Once, at progression or death from any cause
  PFS from the date of the next treatment to disease progression or death from any cause
Overall survival (OS) | Once, death from any cause or lost of follow-up
  Time from either the date of diagnosis or the start of treatment for a disease, such as cancer, that patients diagnosed with the disease are still alive

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No